CLINICAL TRIAL: NCT02873468
Title: Randomized, Double-blind, Multicentric, Parallel, National, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Three Doses of Florence Oral Suspension in Adults With Eosinophilic Esophagitis
Brief Title: Efficacy and Safety of Three Doses of Florence Oral Suspension in Adults With Eosinophilic Esophagitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0718 - FLORENCE
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Florence 30 (Experimental)
  Interventions: Drug: Florence 30 μg/mL
- Florence 60 (Experimental)
  Interventions: Drug: Florence 60 μg/mL
- Florence 90 (Experimental)
  Interventions: Drug: Florence 90 μg/mL
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Florence 30 μg/mL — 10 mL, oral, twice a day.
  Other Names: EMS oral suspension
  Arms: Florence 30
Drug: Florence 60 μg/mL — 10 mL, oral, twice a day.
  Other Names: EMS oral suspension
  Arms: Florence 60
Drug: Florence 90 μg/mL — 10 mL, oral, twice a day.
  Other Names: EMS oral suspension
  Arms: Florence 90
Other: Placebo — 10 mL, oral, twice a day.
  Other Names: Florence placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of three doses of Florence oral suspension on changes of eosinophilic infiltration in esophageal biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent;
* Participants aged 18 years or more;
* Participants diagnosed with eosinophilic esophagitis, defined as:

  1. Presence of symptoms of esophageal dysfunction intermittently or continuously during previous week to the screening visit;
  2. Eosinophilic esophageal inflammation with ≥ 15 eosinophils/high-power field, in the screening endoscopy;
  3. Exclusion of other causes of esophageal eosinophilia.

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* Participants with a stricture on endoscopy that prevents passage of the endoscope;
* History of alcohol abuse or drug use;
* Use of concomitant therapies for any reason that may affect the assessment;
* History of gastroesophageal surgery;
* History of the abnormal gastrointestinal disorder;
* Another disorder that causes esophageal eosinophilia;
* Pregnancy or risk of pregnancy and lactating patients;
* Participants with known allergy, contraindication or hypersensitivity to the components of the medicine used in the clinical trial;
* Participation in clinical trial in the year prior to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants presenting a histological response, defined as the presence of ≤ 6 eosinophils/high-power field, at the end of treatment. | 100 days

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study. | 170 days

CONTACTS AND LOCATIONS:
Locations (1):
- Allergisa, Campinas, São Paulo, Brazil